CLINICAL TRIAL: NCT06778642
Title: Comparison of the Postoperative Analgesic Effectiveness of Serratus Posterior Superior Intercostal Plane Block and Serratus Anterior Plane Block in Video-Assisted Thoracoscopic Surgery (VATS)
Brief Title: Postoperative Analgesic Comparison of SPSI Block and SAP Block in Video-Assisted Thoracoscopic Surgery (VATS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Rabia Bayraktar Cabuk, Resident Doctor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UU-AN-RBC-01
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Acute Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The study will include patients aged 18-80 years scheduled for VATS at Uludağ University Medical Faculty Hospital. Patients with ASA I, II, and III classifications will be included.
  Patients will be randomized into two groups:
  Group 1: SPSIPB Group 2: SAPB
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers and participants will be double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Posterior Superior Intercostal Plane Block Group (Active Comparator): In this group, the ultrasound device with a linear probe (38 mm, 6 MHz) will be used. The upper medial border of the scapula on the side of the planned surgery will be identified between the 2nd and 7th ribs. A block needle will be inserted medially to the scapula, advancing into the plane between the serratus posterior superior muscle and the intercostal muscles. A total of 30 ml of 0.25% bupivacaine will be injected, with a maximum dose of 2 mg/kg/day. In other words, the injection will be applied under the SPS muscle, between the rib and the SPS muscle.
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block
- Serratus Anterior Plane Block Group (Active Comparator): In this group, the ultrasound device with a linear probe (38 mm, 6 MHz) will be used. The probe will be placed between the anterior and posterior axillary lines, on the side of the planned surgery, between the 2nd and 7th ribs. The block needle will be advanced to the surface or deeper part of the serratus anterior muscle, into the fascial plane. A total of 30 ml of 0.25% bupivacaine will be injected, with a maximum dose of 2 mg/kg/day, underneath the serratus anterior muscle.
  Interventions: Procedure: Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Serratus Posterior Superior Intercostal Plane Block — Patients undergoing Video-Assisted Thoracoscopic Surgery (VATS) will receive either a Serratus Posterior Superior Intercostal Plane Block (SPSIPB) with bupivacaine after induction and before the surgical procedure begins.
  Arms: Serratus Posterior Superior Intercostal Plane Block Group
Procedure: Serratus Anterior Plane Block — Patients undergoing Video-Assisted Thoracoscopic Surgery (VATS) will receive either a Serratus Anterior Plane Block (SAPB) with bupivacaine after induction and before the surgical procedure begins.
  Arms: Serratus Anterior Plane Block Group

SUMMARY:
In our study, we primarily aimed to compare the postoperative analgesic effectiveness of the Serratus Posterior Superior Intercostal Plane Block and the Serratus Anterior Plane Block, both routinely applied in patients undergoing Video-Assisted Thoracoscopic Surgery (VATS)

DETAILED DESCRIPTION:
In Video-Assisted Thoracoscopic Surgery (VATS), the thoracic cavity is visualized through a small incision in the chest wall. VATS allows for procedures such as lobectomy, bullectomy, and wedge resection. Compared to thoracotomy, VATS offers lower costs, better pulmonary function, less pain, and earlier postoperative mobilization. The success of postoperative rehabilitation in thoracic surgery patients can be improved with minimally invasive procedures and effective pain control.

The multimodal analgesic approach, which involves the combined use of analgesic drugs with different mechanisms (NSAIDs, paracetamol, opioids, etc.) along with regional/local techniques, aims to achieve additive and synergistic effects. This approach reduces the need for high doses of a single analgesic, minimizes side effects, and provides more effective pain control.

Investigators routinely apply opioids, NSAIDs, paracetamol, intravenous patient-controlled analgesia (PCA) devices, and regional techniques such as thoracic paravertebral block, serratus anterior plane block (SAPB), serratus posterior superior intercostal plane block (SPSIPB), and erector spinae plane (ESP) block for postoperative pain management in VATS patients.

The primary objective of this study is to compare the effects of Serratus Posterior Superior Intercostal Plane Block (SPSIPB) and Serratus Anterior Plane Block (SAPB), both routinely used in thoracic anesthesia practice, on postoperative pain scores and analgesic needs in VATS patients.

The SAPB, which is an essential component of multimodal analgesia in thoracic surgery, offers safe and precise analgesic effects with low complication rates. The block covers most VATS incisions and chest tube sites, providing better postoperative analgesia and potentially improving lung function. Similarly, SPSIPB, another thoracic wall fascial plane block, has been shown to be effective in managing both acute and chronic pain. It is reported to provide good analgesia in the thoracic region after VATS.

The study will include patients aged 18-80 years scheduled for VATS at Uludağ University Medical Faculty Hospital. Patients with ASA I, II, and III classifications will be included.

Patients will be randomized into two groups:

Group 1: SPSIPB (n=45) Group 2: SAPB (n=45) Both blocks will be applied after standard anesthesia induction, intubation, surgical positioning, and before surgical incision.

During the intraoperative period, if heart rate or mean arterial pressure (MAP) increases by more than 20% from baseline measurements, IV fentanyl (1 µg/kg) will be administered as needed. Prior to the surgical incision, all patients will receive IV paracetamol (10 mg/kg), tenoxicam (20 mg), and metoclopramide (10 mg) as part of routine practice.

Fifteen minutes before awakening, a patient-controlled analgesia (PCA) device will be connected to each patient. The PCA device will be prepared with 1 mg/ml morphine solution, with a bolus dose of 2 ml and a lockout interval of 15 minutes. In patients with an NRS score of ≥4, IV tramadol (100 mg/2 ml) will be administered as a rescue analgesic. The pain score at the time of rescue analgesia, the time of the first PCA request, and the NRS score at that time will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years undergoing Video-Assisted Thoracoscopic Surgery (VATS)
* Scheduled at Uludağ University Faculty of Medicine Hospital Operating Room
* Classified as ASA I, II, or III according to the American Society of Anesthesiologists (ASA) criteria

Exclusion Criteria:

* Allergy to local anesthetics or contraindications to bupivacaine
* Known or suspected coagulopathy
* Infection at the injection site
* History of thoracic surgery
* Severe neurological or psychiatric disorders
* Severe cardiovascular disease
* Liver failure
* Renal failure (glomerular filtration rate < 15 ml/min/1.73 m²)
* Chronic opioid use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NRS) | 2 days
  Numerical Rating Scale (NRS) The Numerical Rating Scale (NRS) is a commonly used pain assessment tool that allows patients to rate their pain intensity on a scale from 0 to 10.
  0 indicates no pain. 10 indicates the worst possible pain. Patients are asked to choose a number that best represents their pain level at the time of assessment.